CLINICAL TRIAL: NCT05382481
Title: Effect of Anti Xa Monitoring Low Molecular Weight Heparin (LMWH) on Prevention of Venous Thromboembolism in Critically Ill Patients：A Randomized Controlled Trial
Brief Title: Anti Xa Monitoring Low Molecular Weight Heparin on Prevention of Venous Thromboembolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-2-2016
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboemboism; low molecular weight heparins; critically ill patients; anti-Xa; randomized controlled trial
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peak value anti-Xa group (Group A) (Experimental): The peak value of anti-Xa level of this group should be remain 0.3～0.5IU/mL. This group will receive low molecular weight heparins (LMWH) 40mg, once a day for the first 3 days. And detect the peak level of anti-Xa after 4 to 6 hours after injection of the third dose of LMWH. Adjust the dose of LMWH according to the peak value of anti Xa.
  Interventions: Diagnostic Test: Peak value anti-Xa
- Trough value anti-Xa group (Group B) (Experimental): The trough value of anti-Xa level of this group should be remain 0.1～0.2IU/mL. This group will receive low molecular weight heparins (LMWH) 40mg, once a day for the first 3 days. And detect the trough level of anti-Xa after 12 hours after injection of the third dose of LMWH. Adjust the dose of LMWH according to the trough value of anti Xa.
  Interventions: Diagnostic Test: Trough value anti-Xa
- Control group （Group C） (Placebo Comparator): The control group will not detect the value of anti Xa and not adjust the dose of LMWH.
  This group will receive fixed dose of low molecular weight heparins (LMWH) 40mg, once a day.
  Interventions: Diagnostic Test: Control Group

INTERVENTIONS:
Diagnostic Test: Peak value anti-Xa — This group will receive low molecular weight heparins (LMWH) 40mg, once a day for the first 3 days. And detect the peak level of anti-Xa after 4 to 6 hours after injection of the third dose of LMWH. Adjust the dose of LMWH according to the peak value of anti Xa.
  Arms: Peak value anti-Xa group (Group A)
Diagnostic Test: Trough value anti-Xa — This group will receive low molecular weight heparins (LMWH) 40mg, once a day for the first 3 days. And detect the trough level of anti-Xa after 12 hours after injection of the third dose of LMWH. Adjust the dose of LMWH according to the trough value of anti Xa.
  Arms: Trough value anti-Xa group (Group B)
Diagnostic Test: Control Group — This group will receive fixed dose of low molecular weight heparins (LMWH) 40mg, once a day. And will not detect the level of anti-Xa
  Arms: Control group （Group C）

SUMMARY:
Venous thromboembolism (VTE), which includes deep vein thrombosis (DVT) and pulmonary embolism, is a common cardiovascular disease associated with significant morbidity ranging from painful leg swelling, chest pain, shortness of breath, and even death. About 50% of all VTE events occur as a result of a current or recent hospital admission for surgery or acute medical illness. Hospital-acquired VTE is preventable, with interventions including anticoagulants and mechanical measures, including compression stockings and intermittent pneumatic compression. Prevented hospital acquired VTE is the focus of health services and the strongest hospital strategy to improve patient health in the world.

DETAILED DESCRIPTION:
Low molecular weight heparins (LMWH) are commonly used injectable anticoagulants for venous thromboembolism (VTE) prophylaxis and treatment. LMWH forms an inhibitory complex with antithrombin to inactivate activated factor X (Xa). Due to the predictable pharmacokinetics and pharmacodynamics of LMWH, it is not necessary to routinely monitor anti-Xa levels. However, LMWH pharmacokinetics and pharmacodynamics may be less predictable in certain patient populations including renal impairment, obesity, malignancy, or pregnancy .

Both increased risk of bleeding and suboptimal efficacy are possible in obese patients. LMWHs distribute into lean body mass, therefore, obese patients with a lower proportion of lean body mass to adipose tissue receiving LMWH dosed according to actual body weight may achieve supratherapeutic drug concentrations which could increase bleeding risk . On the other hand, fixed-dose VTE prophylaxis regimens do not account for higher body weight associated with obesity potentially resulting in subtherapeutic drug concentrations increasing the risk for therapeutic failure.

As LMWH are primarily renally eliminated, impaired renal function can contribute to drug accumulation and increased risk of major bleeding.The prolonged LMWH monotherapy used in cancer-associated VTE treatment also raises concerns about drug accumulation and increased bleeding, especially in those with fluctuating renal function. In addition, pregnancy can potentially increase the clearance and volume of distribution of LMWH, increasing the potential for subtherapeutic anti-Xa levels. Thus, anti-Xa level assays are often performed for these specific patient populations in an attempt to provide optimal LMWH therapy.

Critically ill patients are higher risk populations of VTE and bleeding with complex conditions, for example sedation, mechanical ventilation, central venous catheter, and have severe infection, renal insufficiency/failure. So, the purpose of this RCT is to explore the effect of anti Xa monitoring LMWH in preventing VTE in critically ill patients and the optimal time of anti Xa monitoring, reduce mortality and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* No gender limited
* Prospectively screened for risk and included if they received LMWH
* The patient or his / her legal representative is able and willing to sign the informed consent

Exclusion Criteria:

* History of hemorrhage or high risk of hemorrhage, including subarachnoid hemorrhage, cerebral hemorrhage, traumatic brain injury, blood system diseases, etc
* Severe renal insufficiency before randomization (creatinine clearance rate (CCr) < 30mL/min)
* Expected length of ICU stay less than 3 days
* Known to be allergic to LMWH
* Pregnancy
* History of heparin induced thrombocytopenia
* Patients with iliac vein compression syndrome
* Receive non LMWH for prevention VTE according to the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 858 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
number of VTE | 14 days after randomization
  VTE include symptomatic VTE or asymptomatic VTE at day 14

SECONDARY OUTCOMES:
number of targets reached of peak value or trough value of anti Xa for the first time | 14 days after randomization
  LMWH 40mg，once a day, 3 day later, the peak value or trough value of anti Xa for the first time
number of hemorrhage | 14 days after randomization
  Major hemorrhage include 1)symptomatic hemorrhage in a major organ such as intracranial hemorrhage, intra spinal, intraocular, retro peritoneal, intra-articular, pericardial and muscle bleeding causing a compartment syndrome; 2)symptomatic hemorrhage causing a fall in hemoglobin of at least 2 g / dL or leading to a transfusion of at least two blood unit.
number of all cause in-hospital death | 14 days and in hospital
  Cause and date of death

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang C, Ning YC, Song LP, Li PJ, Wang FH, Ding MX, Jiang L, Wang M, Pei QQ, Hu SM, Wang H. Anti-factor Xa level monitoring of low-molecular-weight heparin for prevention of venous thromboembolism in critically ill patients (AXaLPE): protocol of a randomised, open-label controlled clinical trial. BMJ Open. 2023 Oct 25;13(10):e069742. doi: 10.1136/bmjopen-2022-069742. PMID 37880168